CLINICAL TRIAL: NCT04102423
Title: Investigation of the Natural Progression of Clonal Hematopoiesis of Indeterminate Potential and Clonal Cytopenia of Undetermined Significance.
Brief Title: CHIP/CCUS Natural History Protocol
Status: Recruiting | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190139; 19-H-0139
Record Dates: First submitted 2019-09-24; First posted 2019-09-25 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01-26

CONDITIONS: Clonal Hematopoiesis of Indeterminate Potential; Clonal Cytopenia of Undetermined Significance
Keywords: Cytopenia; Myelodysplastic Syndrome; Somatic Mutations; Natural History
MeSH Terms: conditions — Cytopenia; Myelodysplastic Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CCUS: All participants meeting the criteria for CCUS
- CHIP: Subjects will be split into five cohorts depending on specific mutations

SUMMARY:
Background:

Clonal Hematopoiesis of Indeterminate Potential (CHIP) is a change in a person s DNA that can increase a person s risk of developing blood cancers or cardiovascular disease. CHIP occurs mostly occurs in older people. Clonal cytopenia of undetermined significance (CCUS) occurs when one or more blood cell types is lower than it should be and is associated with a change in their DNA. Researchers want to learn more about how CHIP and CCUS progress.

Objective:

To examine the natural history of people in a study of CHIP and CCUS to (1) verify the association of myeloid somatic mutations with atherosclerosis and blood cancers, and (2) find new potential clinical associations.

Eligibility:

Adults 18 and older with CHIP with a somatic pathogenic variant associated with blood cancers. Adults with CCUS are also needed.

Design:

Potential participants will be screened with gene testing. For this, they will give a blood sample. They will also be enrolled in NHLBI screening protocol #97-H-0041. Those who pass this screening will visit the NIH Clinical Center for more screening tests. For this, they will give a blood sample. They will have a physical exam. They will give their medical history. They may give a urine sample. Those with CCUS will have bone marrow taken.

Eligible participants will give blood and urine samples. Their heart activity will be monitored and tested. The arteries in their neck will be assessed using ultrasound. They will have liver and heart scans. They will have a bone mineral density scan. They will have lung function tests. They will have the inside of their cheek swabbed or have a skin punch biopsy. They will have the option to have advanced scans done of their heart and full body but this is not required.

Participants will have yearly follow-up visits for 10 years. They will repeat the above procedures every 1-3 years depending on the procedure.

DETAILED DESCRIPTION:
Clonal Hematopoiesis of Indeterminate Potential (CHIP) has been defined as the presence of a somatic pathogenic variant associated with hematological malignancy, with an allele fraction of at least 2%, without morphological evidence of bone marrow dysplasia or neoplasia. Such variants are small, occur in leukocytes and are found in a substantial proportion of the healthy aging population using next generation sequencing (NGS). They are thought to represent a pre-neoplastic phase of hematological malignancy, particularly myeloid disorders such as myelodysplastic syndromes (MDS) and acute myeloid leukemia (AML). They are considered by some to be analogous to monoclonal B cell lymphocytosis (MBL), or monoclonal gammopathy of uncertain significance (MGUS) as precursors for chronic lymphocytic leukemia (CLL) and myeloma respectively, and, with a similar rate of progression of 0.5%-1% per year.

CHIP is strongly associated with advancing age with a prevalence of up to 10% in those >65 years of age compared to 1% in those <50 years of age, and has also been associated with an increased atherosclerotic risk, and an increase in overall mortality. Despite this association, most people with CHIP are denoted healthy and do not progress to hematological malignancy. Those with low blood counts in association with a - termed clonal cytopenias of undetermined significance (CCUS) - do show a significantly higher rate of progression to myeloid malignancy, more analogous to patients with low risk MDS, though they are currently not classified as such as they lack the morphological dysplasia or defining chromosomal abnormalities.

The optimal follow-up and management of CHIP and CCUS is not yet established - evidence has suggested that factors such as which specific variant, how many variants are present, and the frequency at which these variants increase can help us to delineate high and low risk status. Some recent data has shown that the presence of CHIP is associated with increased levels of inflammation. In depth, investigation should provide further insight into the pathogenesis and progression of this process. The establishment of a natural history protocol will allow patients with CHIP and CCUS to be followed prospectively in a clinical setting. This protocol will have many collaborators from different institutes providing expertise including National Human Genome Research Institute (NHGRI), National Heart, Lung and Blood Institute (NHLBI), National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK), and the Department of Laboratory Medicine (DLM).

ELIGIBILITY:
* Participants with Clonal Hematopoiesis of Indeterminate Significance (CHIP):

INCLUSION CRITERIA:

* Greater than or equal to 18 years of age
* Willingness and capacity to provide written informed consent
* Presence of a somatic pathogenic variant associated with hematological malignancy
* Variant allele fraction of greater than or equal to 2% in at least one identified somatic pathogenic variant

EXCLUSION CRITERIA:

* Known diagnosis of a hematological malignancy or bone marrow failure syndrome (excluding MGUS or MBL)
* Presence of a cytopenia:

  --Hemoglobin, <10 g/dL; platelet count, <100 X 10^9 /L; or absolute neutrophil count, <1.5 X 10^9 /L
* Pregnant at the time of recruitment

Participants with Clonal Cytopenia of Uncertain Significance (CCUS):

INCLUSION CRITERIA:

* Greater than 18 years of age
* Willingness and capacity to provide written informed consent
* Presence of a somatic pathogenic variant associated with hematological malignancy without morphological evidence of

myelodysplasia and without a MDS defining cytogenetic abnormality

* Variant allele fraction of greater than or equal to 2% in at least one identified somatic pathogenic variant
* Bone marrow aspirate and biopsy excluding hematological malignancy and MDS
* Presence of a cytopenia for >30 days

  * Hemoglobin, <10 g/dL; platelet count, <100 X10^9 /L; or absolute neutrophil count, <1.5 X10^9 /L
  * At least 2 CBCs documented in a non-hospitalized patient at least 3 days apart

EXCLUSION CRITERIA:

* Known diagnosis of a hematological malignancy or bone marrow failure syndrome (excluding MGUS or MBL)
* Morphological evidence of dysplasia on bone marrow aspirate / biopsy 10% dysplastic cells in any hematopoietic lineage
* Ringed sideroblasts >15%
* Presence of MDS defining cytogenetic abnormality

  * del(7q)
  * del(5q)
  * 17q or t(17p)
  * del(13q)
  * del(11q)
  * del(12p) or t(12p)
  * del(9q)
  * idic(X)(q13)
  * t(11;16)
  * t(3;21)
  * t(1;3)
  * t(2;11)
  * inv(3)/t(3;3)
* t(6;9)

  --Note: As a sole cytogenetic abnormality in the absence of morphological criteria, gain of chromosome 8, del(20q) and loss of chromosome Y are not considered definitive evidence of MDS.
* Alternate hematological diagnosis causing cytopenia
* Pregnant at time of recruitment
* Previous chemotherapy or radiotherapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary Clinical
Sampling Method: Non-Probability Sample
Enrollment: 306 (Estimated)
Dates: Start 2020-03-03 (Actual); Primary Completion 2033-09-15 (Estimated); Study Completion 2033-09-15 (Estimated)

PRIMARY OUTCOMES:
Verify the previously studied association of myeloid somatic mutations with hematological malignancy | 10 years
  Association of myeloid somatic mutations with hematological malignancy
Verify the previously studied association of myeloid somatic mutations with atherosclerosis | 10 years
  Association of myeloid somatic mutations with atherosclerosis
Immune response | 10 years
  Assessing immune response by measuring markers of inflammation
Examine potential new clinical associations | 10 years
  New clinical associations
Development of cytopenia, hematological malignancy, and the size and stability of leucocyte somatic mutations | 10 years
  Cytopenia, hematological malignancy, and the size and stability of leucocyte somatic mutations

SECONDARY OUTCOMES:
Relationship between CHIP/CCUS and chronic viral infections such as CMV, EBV, HSV, HIV, Hepatitis B and Hepatitis C | 10 years
  To establish whether there is a relationship between CHIP/CCUS and chronic viral infections such as CMV, EBV, HSV, HIV, Hepatitis B and Hepatitis C
Relationship between CHIP/CCUS and atherosclerosis, diabetes, and metabolic syndrome | 10 years
  To establish whether there is a relationship between CHIP/CCUS and atherosclerosis, diabetes, and metabolic syndrome
Correlation between CHIP/CCUS and vitamin levels | 10 years
  To establish whether there is a correlation between CHIP/CCUS and vitamin levels
Correlation between CHIP/CCUS and chronic renal impairment | 10 years
  To establish whether there is a correlation between CHIP/CCUS and chronic renal impairment
Correlation between CHIP/CCUS and chronic lung disease | 10 years
  To establish whether there is a correlation between CHIP/CCUS and chronic lung disease
Correlation between CHIP/CCUS and chronic liver disease | 10 years
  To establish whether there is a correlation between CHIP/CCUS and chronic liver disease

CONTACTS AND LOCATIONS:
Overall Officials: Emma M Groarke, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-H-0139.html